CLINICAL TRIAL: NCT04670523
Title: Early Postoperative Day 0 Chest Tube Removal After Thoracoscopic Minor Surgeries. A Randomized Controlled Clinical Trial.
Brief Title: Early Postoperative Day 0 Chest Tube Removal After Thoracoscopic Minor Surgeries
Acronym: CTremoval
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EROCT
Record Dates: First submitted 2020-11-27; First posted 2020-12-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Lung Pathologies of Unclear Etiology

STUDY DESIGN:
Intervention Model Description: Prospective randomization of patients after minor thoracic operations into two different groups. The patients of the study group are getting their chest tube removed according to our current airleak protocol (Flow <20 mL/ min on digital suction device) but already in the operating room after wound closure. If airleak is persisting than chest tube removal will be performed according to the traditional protocol not earlier than on postoperative day 1. In the control group, the chest tube gets removed according to the investigators' traditional standard protocol not earlier than on postoperative day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Other): Test group: The patients of the study group are getting their chest tube removed according to the investigators' current airleak protocol (Flow <20 mL/ min on digital suction device) but already in the operating room immediately following wound closure (Postoperative day 0 (POD0)). If airleak is persisting than chest tube removal will be performed according to the traditional protocol not earlier than on postoperative day 1 (POD 1).
  Interventions: Procedure: Early postoperative day 0 (POD 0) chest tube removal.
- Control group (Other): In the control group, the chest tube gets removed according to the investigators' traditional standard protocol not earlier than on postoperative day 1 (POD1).
  Interventions: Procedure: Chest tube removal according to traditional standard protocol not earlier than on postoperative day 1 (POD 1).

INTERVENTIONS:
Procedure: Early postoperative day 0 (POD 0) chest tube removal. — Chest tube removal is a standard bedside intervention after lung resections. Its time point is normally defined according a traditional standard airleak threshold. Traditionally, in our department this threshold will be respected not earlier than 1 day after the operation. The patients of the study group are getting their chest tube removed according to our current airleak protocol (Flow <20 mL/ min on digital suction device) but already in the operating room after wound closure (POD 0). If airleak is persisting than chest tube removal will be performed according to the traditional protocol not earlier than on postoperative day 1 (POD 1).
  Arms: Test group
Procedure: Chest tube removal according to traditional standard protocol not earlier than on postoperative day 1 (POD 1). — Chest tube removal according to traditional standard protocol not earlier than on postoperative day 1 (POD 1).
  Arms: Control group

SUMMARY:
The safe conditions for early chest tube removal have been progressively questioned and redefined around reliable digital air flow criteria and extension of liquid threshold accepted. Nevertheless, in current practice, the chest tube remains in restricting early mobilization and optimal compliance with ERAS programme, during the first crucial 24 h after surgery. Thus, to go further, the investigators decide to assess in this study the safety of POD 0 chest tube removal after minor thoracic operations in patients in health condition tolerating operation and anesthesia.

DETAILED DESCRIPTION:
Chest tube management is a key element of postoperative care after thoracic surgeries for different indications. During the last decade, minimally invasive surgery and enhanced recovery after surgery (ERAS) programmes have radically changed the equation of recovery, contributing to reduce postoperative morbidity and enhance quality of life, but the chest tube remains its Achilles heel, still providing postoperative pain and impairing pulmonary function. In this view, early chest tube removal has been widely promoted not only for its economic benefits on length of stay but also for improving quality of life and potentially reducing postoperative complications. In parallel, the change from traditional chest drainage devices to electronic devices has also enabled a more accurate air leak measurement with reduction of interobserver variability, decreased chest drainage duration and shortened LOS. The safe conditions for early chest tube removal have been progressively questioned and redefined around reliable digital air flow criteria and extension of liquid threshold accepted. Nevertheless, in current practice, the chest tube remains in restricting early mobilization and optimal compliance with ERAS programme, during the first crucial 24 h after surgery. Thus, to go further, the investigators decide to assess in this study the safety of POD 0 chest tube removal after minor thoracic operations in patients in health condition tolerating operation and anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Thoracoscopic extra-anatomical lung resection (surgical lung biopsy)
2. Thoracoscopic pleural biopsy
3. Signed consent
4. Age of majority

Exclusion Criteria:

1. Anatomical resection
2. Empyema
3. Pleural effusion
4. Pleurodesis
5. Vulnerable persons (Pregnant women, Children and adolescents)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Pneumothorax requiring chest tube reinsertion | Pneumothorax 2 hours after chest tube removal between postoperative day 0 and 30 (POD 0 - 30)
  Number of patients with pneumothorax requiring chest tube reinsertion after removal of initial chest tube
2. Pleural effusion requiring thoracocentesis | Pleural effusion 2 hours after chest tube removal between POD 0 and 30
  Number of patients with pleural effusion requiring thoracocentesis after removal of first chest tube
3. Prolonged air leak > 5 days | Chest tube removal between POD 6 and 30
  Number of patients with persisting air leak longer than 5 days
4. Re-admission or reoperation due to pleural complication | Up to 1 month after first operation
  Number of patients re-admitted to a hospital after first hospitalization

SECONDARY OUTCOMES:
1. Cardiopulmonary complications (Pneumonia, Atrial fibrillation, ARDS) | Up to 1 month after initial operation
  Number of patients with cardiopulmonary complications (Pneumonia, Atrial fibrillation, ARDS) after operation
2. Re-operation | Up to 1 month after initial operation
  Number of patients requiring a re-operation after initial operation
3. Length of drainage (days) | Up to 1 month after initial operation
  Average of time with chest tube in site
4. Length of stay (days) | Up to 1 month after initial operation
  Average of time in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dorn, PD, Study Director — Chief, Department of General Thoracic Surgery, Inselspital
Locations (1):
- University Hospital of Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be included in a manuscript and published in a journal to share the data and results of the study